CLINICAL TRIAL: NCT05158387
Title: A Phase III, Multicentre, Randomised, Double-blind, Chronic-dosing, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy and Safety of Two Dose Regimens of Tozorakimab in Participants With Symptomatic Chronic Obstructive Pulmonary Disease (COPD) With a History of COPD Exacerbations (TITANIA)
Brief Title: Efficacy and Safety of Tozorakimab in Symptomatic Chronic Obstructive Pulmonary Disease With a History of Exacerbations.
Acronym: TITANIA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D9180C00004; 2021-003771-34 (EudraCT Number)
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; COPD; tozorakimab; exacerbations; ICS; LABA/LAMA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: unblinded administrator/pharmacist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tozorakimab Dose 1 (Experimental): Dosing subcutaneously tozorakimab Dose 1 and placebo
  Interventions: Drug: Tozorakimab
- Tozorakimab Dose 2 (Experimental): Dosing subcutaneously tozorakimab Dose 2
  Interventions: Drug: Tozorakimab
- Placebo (Placebo Comparator): Dosing subcutaneously with equivalent volume to tozorakimab
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tozorakimab — Administered subcutaneously tozorakimab Dose 1 and placebo through Week 52.
  Arms: Tozorakimab Dose 1
Drug: Tozorakimab — Administered subcutaneously tozorakimab Dose 2 through Week 52.
  Arms: Tozorakimab Dose 2
Drug: Placebo — Placebo administered subcutaneously, equivalent volume to tozorakimab through week 52.
  Arms: Placebo

SUMMARY:
The purpose of this Phase III study is to evaluate the efficacy and safety of tozorakimab Dose 1 and Dose 2 administered subcutaneously (SC) in adult participants with symptomatic COPD and history of ≥ 2 moderate or ≥ 1 severe exacerbation of COPD in the previous 12 months. Participants should be receiving optimised treatment with maintenance inhaled therapy (ICS/LABA/LAMA triple therapy, or dual therapy if triple is not considered appropriate) in stable doses throughout at least 3 months prior to enrolment.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 40 years of age and capable of giving signed informed consent.
2. Documented diagnosis of COPD for at least one year prior to enrolment.
3. Post BD FEV1/FVC < 0.70 and post-BD FEV1 >20% of predicted normal value.
4. Documented history of ≥ 2 moderate or ≥ 1 severe COPD exacerbations within 12 months prior to enrolment.
5. Documented optimized inhaled dual or triple therapy at a stable dose for at least 3 months prior to enrolment.
6. Smoking history of ≥ 10 pack-years.
7. CAT total score ≥10, with each of the phlegm (sputum) and cough items with a score ≥ 2

Exclusion Criteria:

1. Clinically important pulmonary disease other than COPD.
2. Radiological findings suggestive of a respiratory disease other than COPD that is significantly contributing to the participant's respiratory symptoms.
3. Current diagnosis of asthma, prior history of asthma, or asthma-COPD overlap. Childhood history of asthma is allowed and defined as asthma diagnosed and resolved before the age of 18.
4. Any unstable disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric disorder, major physical and/or cognitive impairment that could affect safety, study findings or participants ability to complete the study.
5. COPD exacerbation, within 2 weeks prior to randomization, that was treated with systemic corticosteroids and/or antibiotics, and/or led to hospitalization.
6. Active significant infection within the 4 weeks prior to randomization, pneumonia within 6 weeks prior to randomization, or medical condition that predisposes the participant to infection.
7. Suspicion of, or confirmed, ongoing SARS-CoV-2 infection.
8. Significant COVID-19 illness within the 6 months prior to enrolment.
9. Unstable cardiovascular disorder.
10. Diagnosis of cor pulmonale, pulmonary arterial hypertension and/or right ventricular failure.
11. History of known immunodeficiency disorder, including a positive test for HIV-1 or HIV 2.
12. History of positive test or treatment for hepatitis B or hepatitis C (except for cured hepatitis C)
13. Evidence of active liver disease, including jaundice during screening.
14. Malignancy, current or within the past 5 years, except for adequately treated non-invasive basal cell and squamous cell carcinoma of the skin and cervical carcinoma-in-situ treated with apparent success more than one year prior to enrolment. Suspected malignancy or undefined neoplasms.
15. Participants who have evidence of active TB.
16. Participants that have previously received tozorakimab.
17. Any clinically significant abnormal findings in physical examination, vital signs, ECG, or laboratory testing during the screening period, which in the opinion of the investigator may put the participant at risk because of their participation in the study, or may influence the results of the study, or the participant's ability to complete the entire duration of the study.
18. Active vaping of any products or using smoked marijuana within the 6 months prior to randomization and during the study.

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1172 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-01-19 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of moderate to severe COPD exacerbations in participants who are former smokers. | over 52 weeks
  The primary endpoint will be assessed first in the primary population (former smokers with symptomatic COPD and a history of exacerbations, on optimised treatment with maintenance inhaled therapy [triple therapy, or dual therapy if triple is not considered appropriate]) and then assessed in the overall population of participants.

SECONDARY OUTCOMES:
Annualized rate of moderate to severe COPD exacerbations in former or current smokers. | over 52 weeks
  The annualized rate will be assessed in the overall population of participants including current and former smokers with symptomatic COPD and history of exacerbations, on optimised treatment with maintenance inhaled therapy.
Time to first moderate to severe COPD exacerbation in former smokers. | over 52 weeks
  To explore the extent to which treatment with each dose of tozorakimab delays the time to first exacerbation compared with placebo in former smokers.
Mean change from baseline in pre-BD, pre-dose trough FEV1 (mL) in former smokers. | Week 52, or over 52 weeks
  Change from baseline in pre-bronchodilator, pre dose trough FEV1 (mL) in former smokers.
Mean change from baseline in pre-BD, pre-dose trough FEV1 (mL) in the overall population of current and former smokers. | Week 52, or over 52 weeks
  Change from baseline in pre-bronchodilator, pre dose trough FEV1 (mL) in the overall population of current and former smokers.
Percentage of responders achieving MCID in E-RS:COPD total score in former smokers | Week 52
  Responder analyses for E-RS:COPD total score at Week 52 based upon a ≥ 2 point improvement (decrease) from baseline in former smokers.
Percentage of responders achieving MCID in E-RS:COPD total score in the overall population of current and former smokers. | Week 52
  Responder analyses for E-RS:COPD total score at Week 52 based upon a ≥ 2 point improvement (decrease) from baseline in the overall population of current and former smokers.
Mean change from baseline in E-RS:COPD total score in former smokers. | over 52 weeks
  Difference in mean change in E-RS:COPD total score from baseline in former smokers.
Mean change from baseline in E-RS:COPD total score in the overall population of current and former smokers. | over 52 weeks
  Difference in mean change in E-RS:COPD total score from baseline in the overall population of current and former smokers.
Percentage of responders achieving MCID in SGRQ total score in former smokers. | Week 52
  Percentage of participants with a decrease in SGRQ total score of ≥ 4 points from baseline in former smokers.
Percentage of responders achieving MCID in SGRQ total score in the overall population of current and former smokers. | Week 52
  Percentage of participants with a decrease in SGRQ total score of ≥ 4 points from baseline in the overall population of current and former smokers.
Mean change from baseline in SGRQ total score from in former smokers. | over 52 weeks
  Difference in mean change from baseline in SGRQ total score in former smokers.
Mean change from baseline in SGRQ total score from in the overall population of current and former smokers. | over 52 weeks
  Difference in mean change from baseline in SGRQ total score in the overall population of current and former smokers.
Time to first severe COPD exacerbation in former smokers. | over 52 weeks
  To evaluate hazard ratio of first severe COPD exacerbation in former smokers.
Annualized rate of severe COPD exacerbations in former smokers. | over 52 weeks
  The rate ratio of severe COPD exacerbations will be assessed in former smokers.
Change from baseline in CAT total score. | Week 52
  Analyses of change from baseline in CAT total score in former smokers.
Percentage of participants with a decrease in CAT total score in former smokers. | Week 52
  Proportion of participants achieving MCID in CAT total score, a decrease in CAT total score of ≥ 2 points from baseline in former smokers.
Proportion of participants having ≥ 1 healthcare resource utilization type in former smokers. | over 52 weeks
  Proportion of participants having ≥ 1 healthcare resource utilization type in former smokers.
Annualized rate of healthcare resource utilization in former smokers. | over 52 weeks
  Annualized rate of healthcare resource utilization in former smokers.
The change from baseline in mean number of puffs per day in rescue use in former smokers. | over 52 weeks
  Difference in mean number of puffs per day from baseline.
Trough serum concentrations of tozorakimab. | over 52 weeks
  Pharmacokinetics: concentrations of tozorakimab in trough serum.
Presence of anti-drug antibodies. | over 60 weeks
  Immunogenicity: presence of tozorakimab anti-drug antibodies in blood serum.

CONTACTS AND LOCATIONS:
Locations (183):
- United States (34):
  - Research Site, Sheffield, Alabama
  - Research Site, Lincoln, California
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Newark, Delaware
  - Research Site, Bay Pines, Florida
  - Research Site, Cape Coral, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Macon, Georgia
  - Research Site, Greenwood, Indiana
  - Research Site, Bowling Green, Kentucky
  - Research Site, White Marsh, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Buffalo, New York
  - Research Site, The Bronx, New York
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Rock Hill, South Carolina
  - Research Site, Amarillo, Texas
  - Research Site, Boerne, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, McKinney, Texas
  - Research Site, Tomball, Texas
  - Research Site, Webster, Texas
  - Research Site, Williamsburg, Virginia
  - Research Site, Cudahy, Wisconsin
- Australia (9):
  - Research Site, Campbelltown
  - Research Site, Frankstown
  - Research Site, Macquarie University
  - Research Site, Melbourne
  - Research Site, Nedlands
  - Research Site, Southport
  - Research Site, Spearwood
  - Research Site, Wollongong
  - Research Site, Woodville South
- Brazil (8):
  - Research Site, Blumenau
  - Research Site, Botucatu
  - Research Site, Brasília
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Bernardo do Campo
  - Research Site, São Paulo
- Chile (3):
  - Research Site, Curicó
  - Research Site, Santiago
  - Research Site, Talca
- China (33):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changde
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Kunming
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shengyang
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xiamen
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Yinchuan
  - Research Site, Zhanjiang
  - Research Site, Zunyi
- Colombia (4):
  - Research Site, Barranquilla
  - Research Site, Ibagué
  - Research Site, Rionegro
  - Research Site, Zipaquirá
- France (10):
  - Research Site, Brest
  - Research Site, Dijon
  - Research Site, Grenoble
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montivilliers
  - Research Site, Montpellier
  - Research Site, Pessac
  - Research Site, Saint-Herblain
  - Research Site, Toulouse
- Germany (10):
  - Research Site, Ahrensburg
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Darmstadt
  - Research Site, Halle
  - Research Site, Marburg
  - Research Site, München
  - Research Site, München-Pasing
  - Research Site, Peine
- Greece (6):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Exohi Thessaloniki
  - Research Site, Ioannina
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Israel (6):
  - Research Site, Ashkelon
  - Research Site, Beersheba
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Italy (13):
  - Research Site, Bari
  - Research Site, Massa
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Salerno
  - Research Site, San Donà di Piave
  - Research Site, Sassari
  - Research Site, Statte
  - Research Site, Telese Terme
  - Research Site, Tradate
  - Research Site, Vercelli
  - Research Site, Verona
- Research Site, Lima, Peru
- Philippines (3):
  - Research Site, Baguio City
  - Research Site, Cebu City
  - Research Site, Iloilo City
- Poland (13):
  - Research Site, Bialystok
  - Research Site, Bychawa
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Ostróda
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Skierniewice
  - Research Site, Sosnowiec
  - Research Site, Wroclaw
- Research Site, Ponce, Puerto Rico
- Romania (5):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
  - Research Site, Timișoara
- Russia (2):
  - Research Site, Penza
  - Research Site, Saratov
- Taiwan (6):
  - Research Site, Hsinchu
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
  - Research Site, Yunlin
- Thailand (8):
  - Research Site, Bang Kra So
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang,
  - Research Site, Muang
  - Research Site, Mueang
  - Research Site, Nakhon Ratchasima
- United Kingdom (8):
  - Research Site, Bradford
  - Research Site, Corby
  - Research Site, Enfield
  - Research Site, Hampshire
  - Research Site, High Wycombe
  - Research Site, Northwood
  - Research Site, Preston
  - Research Site, Shipley